CLINICAL TRIAL: NCT06423495
Title: Efficacy of Photobiomodulation in the Rehabilitation of Olfactory Dysfunctions Induced by Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaffree & Guinle Universitary Hospital (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Deborah Santos Sales, Deborah Santos Sales, Gaffree & Guinle Universitary Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GaffreeGuinleUH
Record Dates: First submitted 2024-02-22; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Anosmia; Ageusia; COVID-19; Rehabilitation; Laser Therapy
Keywords: Anosmia; ageusia; COVID-19; Rehabilitation; Photobiomodulation
MeSH Terms: conditions — Anosmia; Ageusia; COVID-19

STUDY DESIGN:
Intervention Model Description: The sample will consist of 30 individuals who will be allocated to the low-intensity laser treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low-intensity laser treatment group (Experimental): This is an intervention study. The sample will consist of 30 individuals who will be allocated to the low-intensity laser treatment group.
  Interventions: Device: low-intensity laser treatment

INTERVENTIONS:
Device: low-intensity laser treatment — The experimental group will be subjected to a total of up to 24 sessions (2x a week for up to 12 weeks) of irradiation with red and infrared laser pulsed radiation, with 820mm wavelength, 60w power and 6 energy cages, applied in both nostrils and in 10 points under the tongue.

SUMMARY:
On January 30, 2020, the WHO (World Health Organization) declared the new coronavirus pandemic as the sixth public health emergency of international concern. In February 2020, the virus was designated by the Coronavirus Study Group of the International Committee on Virus Taxonomy as severe acute respiratory syndrome coronavirus 2. Many reports have described the appearance of olfactory or gustatory dysfunction simultaneously with other pre-established symptoms of COVID-19. Symptoms such as loss of taste or smell may appear 2 to 14 days after being infected with COVID-19. Worldwide, evidence regarding anosmia (loss of smell) and dysgeusia (change in taste) has been associated with COVID-19 infection. OBJECTIVES: To evaluate the effectiveness of low-intensity laser in treating changes in smell and taste after COVID-19 infection and map which changes obtained the best results. MATERIAL AND METHODS: This is an intervention study whose sample will consist of 30 individuals with loss of smell and taste for more than 6 months after COVID-19 infection, aged 18 years or older.

DETAILED DESCRIPTION:
objective: To evaluate the effectiveness of low-intensity laser in resolving chemosensory symptoms caused by COVID-19.

This is an intervention study. The sample will consist of 30 individuals who will be allocated to the low-intensity laser treatment group.

The patients will come from research at the COVID-19 outpatient clinic at the Gafree Guinle University Hospital - UNIRIO. Patients who agree to participate in the study will be informed about the objective of the research and will sign an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complained of loss of smell and taste more than 6 months after COVID-19 infection, aged 18 years or older, with proof of infection by PCR, will be included in the study.

Exclusion Criteria:

* Patients with comorbidities prior to COVID-19 infection that could interfere with the functions of smell and taste will be excluded from the study; patients with a history of head and neck cancer, epileptic patients; mouth breathing patients; and pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
effectiveness of low-intensity laser in the treatment of olfactory dysfunction in long term covid-19 | 20 minutes session with photobiomodulation therapy twice a week, for a total of 16 sessions
  evaluate the effectiveness of low-intensity laser

CONTACTS AND LOCATIONS:
Overall Officials: Claudia CF Vasconcelos, PHD, Study Director — federal university of the state of rio de janeiro - UNIRIO; Mariana B Hammerle, MD, Study Chair — University hospital Gafree Guinle - UNIRIO; DEBORAH SANTOS SALES, PHD, Principal Investigator — University hospital Gafree Guinle - UNIRIO
Locations (1):
- university hospital Gafree Guinle, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hammerle MB, Sales DS, Pinheiro PG, Gouvea EG, de Almeida PIFM, de Araujo Davico C, Souza RS, Spedo CT, Nicaretta DH, Alvarenga RMP, Pires KL, Thuler LCS, Vasconcelos CCF. Cognitive Complaints Assessment and Neuropsychiatric Disorders After Mild COVID-19 Infection. Arch Clin Neuropsychol. 2023 Feb 18;38(2):196-204. doi: 10.1093/arclin/acac093. PMID 36464245
- [Result] Vasconcelos CCF, Hammerle MB, Sales DS, Rueda Lopes FC, Pinheiro PG, Gouvea EG, Alves MCDF, Pereira TV, Schmidt SL, Alvarenga RMP, Pires KL. Post-COVID-19 olfactory dysfunction: carbamazepine as a treatment option in a series of cases. J Neurovirol. 2022 Apr;28(2):312-318. doi: 10.1007/s13365-022-01066-3. Epub 2022 Apr 2. PMID 35366736
- See also: Post-COVID-19 Olfactory and Gustatory Dysfunction: Photobiomodulation Therapy as a Treatment Option in a Series of Cases — https://openneurologyjournal.com/VOLUME/17/ELOCATOR/e1874205X2309190/FULLTEXT/